CLINICAL TRIAL: NCT06806462
Title: Biomolecular Markers of Bone Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: META_BONE; RC-2024-2790611 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-11-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Bone Metastasis
Keywords: bone; metastasis; biomolecular profile
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone metastasis (Other): Patients with breast or lung or renal or gastroenteric tract or prostate carcinomas with bone metastases
  Interventions: Genetic: Biomolecular profile of bone metastases

INTERVENTIONS:
Genetic: Biomolecular profile of bone metastases — Describe the biomolecular profile of bone metastases

SUMMARY:
The goal of this clinical trial is to characterize the biomolecular profile of bone metastases to define the predisposing profiles of bone metastasis, in patients with breast or lung or renal carcinomas or of the gastroenteric or prostate tract with bone metastasis.

The main question it aims to answer is:

Is it possible to predict the progression of bone metastasis by identifying biomarkers as risk factors for bone metastasis?

DETAILED DESCRIPTION:
Metastasization is a process that involves molecular change: potentially colonizable healthy tissues, particularly bone marrow, may "respond" to the production of factors released by the primary tumor, changing some of their funcional molecular characteristics in order to facilitate colonization by circulating tumor cells.

This study aims to describe the biomolecular profile of bone metastases. For this purpose, as per normal clinical practice, patients with carcinomas and who have developed bone metastases will undergo sampling of the metastases and primary tumors.

The activities will have multidisciplinary management. The study will include patients with carcinoma with bone metastases for whom the collection of biological material from the primary lesion and/or bone metastasis is an integral part of the diagnostic-therapeutic procedure or patients for whom, by clinical practice, a biopsy collection is performed because:

* histologic evaluation of the primary or metastatic lesion has been requested;
* a pathologic fracture to be treated surgically occurs;
* prophylactic orthopedic stabilization is required.

These samples will later be analyzed from a molecular point of view in order to identify a biomolecular profile that can help in defining profiles predisposing to bone metastasis and profiles predisposing to pathological fracture risk.

Unsupervised analysis of the emerged transcriptomes will be conducted:

1. regardless of tumor histotype (in order to highlight any common facilitating factors for bone metastasis and osteolytic activity),
2. by histotype,
3. by type of metastasis (osteolytic vs osteosclerotic).

To eliminate analysis error and bias, analyses will be conducted on fresh samples from needle biopsy or intraoperative sampling.

Emerging evidence on transcriptomic analysis will be validated with protein analysis methods and compared with evidence alreadỳ available in the literature.

The analysis being conducted for this study does not influence clinical practice, and all procedures are part of normal clinical practice in the management of patients with bone metastases from carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patients with breast or lung or renal or gastroenteric tract or prostate with bone metastases
* Patients who knowingly express willingness to participate in the study after signing the written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Bone metastasis profiling | up to 100 weeks
  Characterizing the biomolecular profile of bone metastasis to define the predisposing profiles of bone metastasis.
  Transcriptional profile of
  * RANK/RANKL
  * OPG
  * PTHLH
  * IL-1/6/7/8/11,
  * TNF-alfa
Fracture pathological profiling | up to 100 weeks
  Characterizing the biomolecular profile of bone metastasis to define the predisposing risk profiles of fracture pathological. Fracture event yes/no and association with primary outcomes.

SECONDARY OUTCOMES:
Comparison between the biomolecular profile of the mestastases and the primary tumor | up to 100 weeks
  Trascriptional profile of:
  * RANK/RANKL,
  * OPG
  * PTHLH
  * IL-1/6/7/8/11
  * TNF-alfa
Comparison between the biomolecular profiles of osteolytic and osteosclerotic metastases | up to 100 weeks
  Trascriptional profile of:
  * RANK/RANKL,
  * OPG
  * PTHLH
  * IL-1/6/7/8/11
  * TNF-alfa
Measuring PTH-rp (parathormone-related peptide) levels and the risk of pathologic facture | Every 3-6 months
  Dosage of PTHrp

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sambri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy